CLINICAL TRIAL: NCT01064908
Title: A Study To Determine The Effectiveness Of A New Oxygen Mask At Increasing Arterial Oxygen Content During Carotid Endarterectomy Under Local Anaesthesia
Brief Title: A New Oxygen Mask for Carotid Endarterectomy Under Local Anaesthesia
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr C. Mark Harper, Consultant Anaesthetist, Brighton and Sussex University Hospitals NHS Trust
Other Study IDs: 09/181/HAR
Record Dates: First submitted 2010-02-04; First posted 2010-02-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Stroke; TIA; Surgery; Anaesthesia; Carotid Stenosis
Keywords: Endarterectomy, Carotid; Carotid stenosis; Oxygen mask
MeSH Terms: conditions — Stroke; Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carotid endarterectomy: Patients who are undergoing elective carotid endarterectomy under local anaesthesia
  Interventions: Device: OxyMask

INTERVENTIONS:
Device: OxyMask — Novel vortex oxygen delivery mask
  Other Names: OxyMask Adult Large

SUMMARY:
The purpose of this study is to determine the effectiveness of oxygenation and patient-acceptability of a novel oxygen face mask in patients undergoing carotid endarterectomies (CEAs).

DETAILED DESCRIPTION:
Carotid endarterectomy (CEA) is a procedure to remove plaques from a carotid artery (one of the two main arteries supplying blood to the brain). The procedure is effective at reducing the risk of subsequent stroke. To access the artery, an incision is made in the artery wall which means that the artery must be clamped in order to prevent blood loss. Consequently, the blood supply (and therefore oxygen supply) to the brain is reduced. To ensure that the patient has sufficient oxygen to avoid brain damage, this procedure is often carried out under local anaesthetic as this means the anaesthetist can talk to them during the operation; by this means they can determine the patient's conscious level and whether or not they need supplementary oxygen.

There are various ways to administer the supplementary oxygen. Most oxygen masks completely cover the mouth and nose which inevitably limits patient-doctor communication. Oxygen is therefore usually administered via nasal tubes. However, the actual level of oxygen taken in by the patient is very hard to measure, and at best is only 40%.

A novel mask with an open design. By creating a 'vortex' of oxygen it can deliver higher concentrations of oxygen to the patient without significantly interfering with doctor-patient communication and, at the same time, improving patient comfort.

We wish to test the efficacy of this mask during CEA and plan to do this by measuring the oxygen content of blood directly using blood samples; we also monitor markers of brain damage which may occur from lack of oxygen. Finally, we will survey the patients as to acceptability of the mask.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Booked for carotid endarterectomy under local anaesthetic
* Competent to consent to inclusion

Exclusion Criteria:

* Patient refusal and inability to provide consent
* Patients who are unable to understand instruction or communicate effectively
* Aged below 16 years
* Decreased conscious level during the period of study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Vascular Surgical Outpatients, booked for CEA under local anaesthetic
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary aim of this study the aim is to determine the effectiveness of the vortex oxygen mask in increasing blood oxygen levels during CEA in the awake patient during carotid clamping. | 0 hours

SECONDARY OUTCOMES:
To determine whether or not increased cerebral oxygen levels are associated with reduced cerebral injury, as measured by biomarkers: neuron-specific enolase and S100B. | 2.5 hours.
A further secondary outcome is to determine whether the mask is acceptable to patients, as recorded by a questionnaire. | Within 24 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Mark Harper, MB BS, Principal Investigator — Brighton and Sussex University Hospitals NHS Trust
Locations (1):
- Royal Sussex County Hospital, Brighton, East Sussex, United Kingdom